CLINICAL TRIAL: NCT00249288
Title: Folate Supplementation in Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Principal Investigator, Donald C. Goff, MD, Director of the Schizophrenia Clinical and Research Program, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2004P-000495
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Results first posted 2014-08-06 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Negative Symptoms; Folate
MeSH Terms: conditions — Schizophrenia | interventions — Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Folate (Experimental): Participants will receive a 2 mg/ day dose of folate, for 12 weeks
  Interventions: Drug: Folate
- Placebo (Placebo Comparator): Participants will receive a 2 mg/ day dose of placebo, for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Folate — Folic acid taken as 2, 1mg capsule daily for 12 weeks
  Other Names: Folate or folic acid
  Arms: Folate
Drug: Placebo — Placebo taken as 2, 1mg capsule daily for 12 weeks
  Arms: Placebo

SUMMARY:
This study aims to examine factors potentially contributing to differences in blood folate, homocysteine or B12 levels between schizophrenia patients, to test the hypothesis that low folate is associated with negative symptoms, and to examine the efficacy of folate supplementation for reducing negative symptoms.

DETAILED DESCRIPTION:
This study is a three-month, placebo-controlled trial of folate 2mg/d in 50 schizophrenia patients who score at least a 3 (moderate or greater severity) on at least one of the SANS global assessment subscales, with the exception of the attention global assessment subscale. The specific aims of this study are:

* To examine factors potentially contributing to differences in blood folate, homocysteine or B12 levels between patients at baseline, including dietary intake and cigarette smoking.
* To test the hypothesis that low folate is associated with negative symptoms by examining correlations between red blood cell folate concentrations and clinical ratings of negative symptoms and by comparing folate concentrations in deficit syndrome versus non-deficit syndrome patients. We will also control for dietary intake cigarettes smoking, gender, and age.
* To examine the efficacy of folate supplementation for reducing negative symptoms

ELIGIBILITY:
Inclusion Criteria:

1. Schizophrenia, any subtype
2. Ages 18-68
3. Male or female
4. A score at least a 3 (moderate or greater severity) on at least one of the SANS global assessment subscales, with the exception of the attention global assessment subscale
5. Stable antipsychotic dose for > 6 weeks
6. Capable of providing informed consent

Exclusion Criteria:

1. Unstable medical illness
2. Substance abuse
3. Megaloblastic anemia
4. Non-english speaking

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2003-12; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald C. Goff, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Hill M, Shannahan K, Jasinski S, Macklin EA, Raeke L, Roffman JL, Goff DC. Folate supplementation in schizophrenia: a possible role for MTHFR genotype. Schizophr Res. 2011 Apr;127(1-3):41-5. doi: 10.1016/j.schres.2010.12.006. Epub 2011 Feb 21. PMID 21334854

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty six participants were enrolled; 38 completed screening and 32 received study drug.
Groups:
- Folate: Participants receiving 2 mg/daily of folate, for 12 weeks
Period: Overall Study
Arm/Group | Folate | Placebo
Started | 19 | 19
Initiated Treatment | 17 | 15
Completed | 14 | 14
Not Completed | 5 | 5
Not completed — Lost to Follow-up | 3 | 3
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received 2 mg/daily of placebo, for 12 weeks
- Folate: Patients underwent a 12 week trial of folate 2 mg/d
- Total: Total of all reporting groups
Arm/Group | Placebo | Folate | Total
Number analyzed (Participants) | 15 | 17 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 17 | 32
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (11.3) | 45.5 (9.6) | 46 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 13 | 13 | 26
Region of Enrollment [Number; unit: participants]
  United States | 15 | 17 | 32

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between Baseline Blood Folate and Smoking Status
Description: Baseline blood folate lab levels are reported by smoking status.
Time Frame: Baseline
Population: 1 past smoker and 1 never smoker are missing RBC folate values. For the present analysis, as opposed to a comparison of treatment groups, folate levels are compared across smoking status.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Groups:
- Current Smoker: Study participants with current smoker status
- Past Smoker: Participants with past smoker status
- Never Smoker: Participants with never smoker status
Arm/Group | Current Smoker | Past Smoker | Never Smoker
Number analyzed (Participants) | 17 | 8 | 7
nanograms per milliliter
  Serum folate, ng/ml | 14.6 (3.3) | 14.6 (5.2) | 14.2 (4.1)
  RBC folate, ng/ml: number analyzed (Participants) | 17 | 7 | 6
  RBC folate, ng/ml | 614 (142) | 542 (122) | 475 (161)

2. Primary Outcome: Correlation Between Baseline Blood Folate and MTHFR Genotype
Description: Baseline blood folate lab levels are reported by MTHFR genotype.
Time Frame: Baseline
Population: One participant with CC genotype is missing RBC folate value. For the present analysis, as opposed to a comparison of treatment groups, folate levels are compared across MTHFR genotype.
Measure: Mean (Standard Deviation); unit: nanograms/mL
Groups:
- CC Genotype: Study participants with MTHFR genotype CC
- T- Genotype: Participants with MTHFR genotype T (T allele carrier)
Arm/Group | CC Genotype | T- Genotype
Number analyzed (Participants) | 13 | 15
nanograms/mL
  Serum folate, ng/ml | 13.3 (3.3) | 15.2 (4.1)
  RBC folate, ng/ml: number analyzed (Participants) | 12 | 15
  RBC folate, ng/ml | 624.8 (143.0) | 542.8 (150.6)

3. Primary Outcome: Correlation Between Baseline Blood Folate Levels and Dietary Intake
Description: Baseline blood folate lab levels and dietary intake levels are reported.
Time Frame: Baseline
Population: All study participants at baseline. For the present analysis, as opposed to a comparison of treatment groups, folate levels are described for all participants at baseline.
Measure: Mean (Standard Deviation); unit: nanograms/mL
Groups:
- Overall: All study participants at baseline
Arm/Group | Overall
Number analyzed (Participants) | 32
nanograms/mL
  Serum folate, ng/ml | 14.5 (3.9)
  RBC folate, ng/ml: number analyzed (Participants) | 30
  RBC folate, ng/ml | 569.3 (148.1)

4. Primary Outcome: Efficacy of Folate Supplementation for Reducing Negative Symptoms as Measured by the SANS Modified Total
Description: The change from baseline to week 12 on the scale for the assessment of negative symptoms (SANS) modified total score. Total SANS scores range from 0-100. The SANS is comprised of 5 sub-scales: Affective Flattening or Blunting (score range 0-35), Alogia (score range 0-20), Avolition-Apathy (score range 0-15), Anhedonia-Asociality (score range 0-20), and Attention (0-10). For each sub-scale, the higher the score the more prominent the negative symptoms were. The total score was computed by adding all the sub-scale total scores. To compute change in scores, baseline scores were subtracted from week 12 scores, resulting in a change score. Lower values signify greater improvement (i.e. week 12 score was lower than baseline score). The SANS modified total score is the SANS total score minus the Attention subscale.
Time Frame: Baseline score vs. week 12 score
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Placebo: Participants will receive a 2 mg/ day dose of placebo, for 12 weeks
  Placebo: Placebo taken by mouth daily as 2, 1mg capsule daily for 12 weeks
Arm/Group | Folate | Placebo
Number analyzed (Participants) | 14 | 14
Units on a scale | -8.5 (7.6) | -9.7 (8.5)

5. Primary Outcome: Correlation Between Baseline Serum B12 Levels and Smoking Status
Description: Baseline serum B12 lab levels are reported by smoking status.
Time Frame: Baseline
Population: For the present analysis, as opposed to a comparison of treatment groups, B12 levels are compared across smoking status.
Measure: Mean (Standard Deviation); unit: picograms per milliliter
Arm/Group | Current Smoker | Past Smoker | Never Smoker
Number analyzed (Participants) | 17 | 8 | 7
picograms per milliliter | 625 (273) | 436 (130) | 574 (160)

6. Primary Outcome: Correlation Between Baseline Homocysteine Levels and Smoking Status
Description: Baseline blood homocysteine lab levels are reported by smoking status.
Time Frame: Baseline
Population: 1 participant who have never smoker status is missing plasma homocysteine values. For the present analysis, as opposed to a comparison of treatment groups, homocysteine levels are compared across smoking status.
Measure: Mean (Standard Deviation); unit: micromoles per liter
Arm/Group | Current Smoker | Past Smoker | Never Smoker
Number analyzed (Participants) | 17 | 8 | 6
micromoles per liter | 9.1 (2.6) | 10.8 (1.6) | 9 (2.5)

7. Primary Outcome: Correlation Between Baseline Blood B12 Levels and MTHFR Genotype
Description: Baseline blood B12 lab levels are reported by MTHFR genotype.
Time Frame: Baseline
Population: For the present analysis, as opposed to a comparison of treatment groups, B12 levels are compared across MTHFR genotype.
Measure: Mean (Standard Deviation); unit: picograms per milliliter
Arm/Group | CC Genotype | T- Genotype
Number analyzed (Participants) | 13 | 15
picograms per milliliter | 605.5 (312.9) | 557.1 (170.1)

8. Primary Outcome: Correlation Between Baseline Blood Homocysteine Levels and MTHFR Genotype
Description: Baseline blood homocysteine lab levels are reported by MTHFR genotype.
Time Frame: Baseline
Population: For the present analysis, as opposed to a comparison of treatment groups, homocystein levels are compared across MTHFR genotype.
Measure: Mean (Standard Deviation); unit: micromoles/liter
Arm/Group | CC Genotype | T- Genotype
Number analyzed (Participants) | 13 | 15
micromoles/liter | 9.4 (2.9) | 9.6 (2.3)

9. Primary Outcome: Correlation Between Baseline Serum B12 Levels and Dietary Intake
Description: Baseline serum B12 lab levels and dietary intake levels are reported.
Time Frame: Baseline
Population: For the present analysis, as opposed to a comparison of treatment groups, B12 levels are described for all baseline participants.
Measure: Mean (Standard Deviation); unit: picograms/mL
Arm/Group | Overall
Number analyzed (Participants) | 32
picograms/mL | 566.6 (231.5)

10. Primary Outcome: Correlation Between Baseline Blood Homocysteine Levels and Dietary Intake
Description: Baseline blood homocysteine lab levels and dietary intake levels are reported.
Time Frame: Baseline
Population: All study participants at baseline. For the present analysis, as opposed to a comparison of treatment groups, homocysteine levels are described for all baseline participants.
Measure: Mean (Standard Deviation); unit: micromoles/liter
Arm/Group | Overall
Number analyzed (Participants) | 31
micromoles/liter | 9.6 (2.4)

11. Primary Outcome: Correlation Between Baseline Blood Folate or B12 Levels and Dietary Intake
Description: Baseline blood folate and B12 lab levels and dietary intake levels are reported.
Time Frame: Baseline
Population: All participants at baseline. For the present analysis, as opposed to a comparison of treatment groups, folate and B12 levels are described for all baseline participants.
Measure: Mean (Standard Deviation); unit: micrograms
Arm/Group | Overall
Number analyzed (Participants) | 16
micrograms
  Total folate, mcg | 531.3 (386.5)
  Dietary folate, mcg | 765.7 (637.7)
  Natural folate, mcg | 198.8 (73.3)
  Synthetic folate, mcg | 333.4 (362.9)
  Total B12, mcg | 7.5 (7.3)

12. Secondary Outcome: Correlations Between Baseline Blood Folate and Clinical Ratings of Negative Symptoms by Comparing Lab Levels in Deficit Syndrome Versus Non-deficit Syndrome Patients
Description: Baseline blood folate lab levels are reported by deficit syndrome status.
Time Frame: Baseline
Population: One deficit syndrome participant and one participant without deficit syndrome are missing RBC folate values. For the present analysis, as opposed to a comparison of treatment groups, folate levels are compared across deficit syndrome status.
Measure: Mean (Standard Deviation); unit: nanograms/mL
Groups:
- Deficit Syndrome: Study participants with deficit syndrome
- Not Deficit Syndrome: Participants without deficit syndrome
Arm/Group | Deficit Syndrome | Not Deficit Syndrome
Number analyzed (Participants) | 17 | 14
nanograms/mL
  Serum folate, ng/ml | 14.9 (4.3) | 14.0 (3.5)
  RBC folate, ng/ml: number analyzed (Participants) | 16 | 13
  RBC folate, ng/ml | 585 (171) | 546 (123)

13. Secondary Outcome: Correlations Between Baseline Blood B12 Levels and Clinical Ratings of Negative Symptoms by Comparing Lab Levels in Deficit Syndrome Versus Non-deficit Syndrome Patients
Description: Baseline blood B12 lab levels are reported by deficit syndrome status.
Time Frame: Baseline
Population: For the present analysis, as opposed to a comparison of treatment groups, B12 levels are compared across deficit syndrome status.
Measure: Mean (Standard Deviation); unit: picograms/mL
Arm/Group | Deficit Syndrome | Not Deficit Syndrome
Number analyzed (Participants) | 17 | 14
picograms/mL | 603 (193) | 513 (275)

14. Secondary Outcome: Correlations Between Baseline Blood Homocysteine Levels and Clinical Ratings of Negative Symptoms by Comparing Lab Levels in Deficit Syndrome Versus Non-deficit Syndrome Patients
Description: Baseline blood homocysteine lab levels are reported by deficit syndrome status.
Time Frame: Baseline
Population: One participant without deficit syndrome is missing homocysteine. For the present analysis, as opposed to a comparison of treatment groups, homocysteine levels are compared across deficit syndrome status.
Measure: Mean (Standard Deviation); unit: micromoles/liter
Arm/Group | Deficit Syndrome | Not Deficit Syndrome
Number analyzed (Participants) | 17 | 13
micromoles/liter | 9.4 (2.6) | 9.7 (2.5)

ADVERSE EVENTS:
Groups:
- Placebo: Participants receiving 2mg/daily of placebo, for 12 weeks
Arm/Group | Folate | Placebo
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No